CLINICAL TRIAL: NCT03373864
Title: Hypobaric Lateral Spinal Anesthesia Versus General Anesthesia: Hemodynamic Stability and Short Term Cardiovascular Complications in Elderly Patients Undergoing Hip Fracture Surgery.
Brief Title: Hypobaric Lateral Spinal Anesthesia Versus General Anesthesia for the Hip Fracture Surgery
Acronym: RACHYP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0513
Record Dates: First submitted 2017-12-07; First posted 2017-12-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hip Fractures
Keywords: Unilateral spinal anesthesia; general anesthesia; hemodynamic stability; MINS; hip fracture; elderly; AKI
MeSH Terms: conditions — Hip Fractures | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral spinal anesthesia (Experimental): In this arm, the patients will have a hypobaric lateral spinal anesthesia. Sedation can be added for the patients comfort.
  Interventions: Procedure: Unilateral spinal anesthesia
- General anesthesia (Active Comparator): In this arm, the patients will have a general anesthesia.
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Unilateral spinal anesthesia — Unilateral spinal anesthesia with hypobaric local anesthesia allowing a lateralized anesthesia of the fractured limb.
  Arms: Unilateral spinal anesthesia
Procedure: General anesthesia — General anesthesia following the latest recommendations for elderly patients (SFAR 2017)
  Arms: General anesthesia

SUMMARY:
Hip fracture is a frequent pathology, involving elderly patients with many co-morbidities ; therefore, post-operative morbidity and mortality is high. It is reported that intra-operative hemodynamics correlate with post-operative complications such as myocardial injury after non-cardiac surgery (MINS) or acute kidney injury (AKI) ; that is why elderly patients undergoing hip fracture surgery should benefit from a better hemodynamic stability.

Low-dose hypobaric lateral spinal anesthesia with a reduced dose of local anesthetic has been shown to have better hemodynamic stability than conventional spinal anesthesia. It has also been reported that general anesthesia and conventional spinal anesthesia in elderly patients undergoing hip fracture surgery have the same hemodynamic effect. However, no published study has compared low-dose hypobaric lateral spinal anesthesia to general anesthesia with regards to hemodynamic effects.

The aim of the present study is to compare the intra-operative hemodynamics of low-dose hypobaric lateral spinal anesthesia with that of general anesthesia in elderly patients undergoing hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

- Every patient aged 70 years or more who undergoes urgent surgery for a traumatic hip fracture.

Exclusion Criteria:

* Patients younger than 70 years of age
* Pathological fractures or multiple trauma
* Contraindications to spinal anesthesia:
* allergy to the local anesthetic
* patients treated by clopidogrel (Plavix®)
* patients treated by oral anticoagulants: dabigatran (Pradaxa®), rivaroxaban (Xarelto®), or apixaban (Eliquis®).
* Coagulation disorders: (Prothrombin Time < 50 %, or Partial Thromboplastin Time ratio > 1.5, or platelets < 80 G/L),
* Local infection of the puncture site
* hyperthermia (> 38.5°C)
* agitated patients
* patients included in another study
* patients under judicial protection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Number of episode of severe intraoperative hypotension | At Day 0
  Occurrence of an episode of severe hypotension defined as a mean arterial pressure (MAP) < 65 mmHg for more than 12 minutes during the operative time.

SECONDARY OUTCOMES:
All-cause mortality | 30 days after surgery
Myocardial injury after non cardiac surgery (MINS) occurence | 3 days after surgery
  Elevated troponin T level (troponin T > 100 ng/L) in aged patients (over 75 years) and for patients under the age of 75 years old Troponin T> 34 ng/L for men and troponin T > 16 ng / L for women, in a blood test performed in the first 3 days after surgery due to a myocardial ischemia.
Acute kidney injury (AKI) occurence | 3 days after surgery
  Postoperative AKI is defined as an increase in serum creatinine between preoperative and postoperative values (increase of more than 1.5-fold or more than 0.3mg/dL of the value before surgery.)
Hemoglobin rate | 1 day after surgery
  Mean decrease between preoperative and postoperative values at 1st and 3rd day after surgery
Hemoglobin rate | 3 days after surgery
  Mean decrease between preoperative and postoperative values at 1st and 3rd day after surgery
Blood loss | At Day 0
  Intraoperative blood loss : quantity of blood in the suction container
Quantity of ephedrine used during the intervention | At Day 0
  Quantity of ephedrine used during operative time and recovery room
Quantity of noradrenaline used during the intervention | At Day 0
  Quantity of noradrenaline used during operative time and recovery room
Number of episodes with a MAP < 65 mmHg for more than 12 minutes during operative time | At Day 0
Total time with MAP < 65 mmHg for more than 12 minutes during operative time | At Day 0
Hospitalisation time | Up to 45 days after surgery
Number of episode of severe hypotension in the recovery room. | At Day 0
  Occurrence of an episode of severe hypotension defined as a mean arterial pressure (MAP) < 65 mmHg for more than 12 minutes in the recovery room.

CONTACTS AND LOCATIONS:
Overall Officials: Claire DELSUC, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot - Service d'Anesthésie-Réanimation, Lyon, France

REFERENCES:
- [Result] Simonin M, Delsuc C, Meuret P, Caruso L, Deleat-Besson R, Lamblin A, Huriaux L, Abraham P, Bidon C, Giai J, Riche B, Rimmele T. Hypobaric Unilateral Spinal Anesthesia Versus General Anesthesia for Hip Fracture Surgery in the Elderly: A Randomized Controlled Trial. Anesth Analg. 2022 Dec 1;135(6):1262-1270. doi: 10.1213/ANE.0000000000006208. Epub 2022 Sep 22. PMID 36135347